CLINICAL TRIAL: NCT07330180
Title: Multicenter, Open-Label, Parallel-Group, Randomized Controlled Study Comparing the Dose-Response Relationship of LED Red Light in Controlling Myopia Progression
Brief Title: Multicenter RCT: LED Red Light Dose-Response in Myopia Progression Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojuan Wang, Director of the Optometry Center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251009041118960
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Myopia, Progressive
Keywords: Myopia; Children; Axial Length; Red-light Therapy
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group A (Experimental): PBM therapy with single intervention duration of 2 minutes + wearing Hoya DIMS defocus lens
  Interventions: Device: Yingtong Vision Rehabilitation Instrument; Device: Hoya DIMS multi-point myopia defocus lens
- Test Group B (Experimental): PBM therapy with single intervention duration of 3 minutes + wearing Hoya DIMS defocus lens
  Interventions: Device: Yingtong Vision Rehabilitation Instrument; Device: Hoya DIMS multi-point myopia defocus lens
- Test Group C (Experimental): PBM therapy with single intervention duration of 4 minutes + wearing Hoya DIMS defocus lens
  Interventions: Device: Yingtong Vision Rehabilitation Instrument; Device: Hoya DIMS multi-point myopia defocus lens
- Control Group D (Active Comparator): Wearing Hoya DIMS defocus lens only
  Interventions: Device: Hoya DIMS multi-point myopia defocus lens

INTERVENTIONS:
Device: Yingtong Vision Rehabilitation Instrument — Input voltage: 6V (4 × 1.5V alkaline dry batteries). Red light wavelength: 650nm; light spot diameter: outer diameter 5.0mm, inner diameter 1.5mm.
  Light source output power: 1.6 mW (±0.1mW at 30mm from the observation window). The Yingtong Vision Rehabilitation Instrument should be used twice a day under the regular communication and supervision of hospital optometrists/coordinators (via phone, WeChat, etc.), with an interval of at least 4 hours.
  Arms: Test Group A; Test Group B; Test Group C
Device: Hoya DIMS multi-point myopia defocus lens — Frame glasses worn on the bridge of the nose

SUMMARY:
The goal of this clinical trial is to verify the effectiveness and safety of non-laser LED red light combined with defocus lens therapy for controlling myopia progression and evaluate the impact of different intervention durations in 6-14 years old children and adolescents with myopia (spherical equivalent refraction: -6.00D ≤ SER ≤ -1.00D), regardless of gender. The main questions it aims to answer are:

[primary hypothesis or outcome measure 1]: Does the combination of Yingtong Vision Rehabilitation Instrument (non-laser LED red light) and Hoya DIMS defocus lens show non-inferior effectiveness to Hoya DIMS defocus lens alone in controlling 6-month axial length change? [primary hypothesis or outcome measure 2]: Do different single intervention durations (2min, 3min, 4min) of non-laser LED red light affect the effectiveness (e.g., axial length change at multiple time points, 12-month SER change) and safety of the combined therapy? If there is a comparison group: Researchers will compare Test Group A (2min PBM therapy + DIMS lenses), Test Group B (3min PBM therapy + DIMS lenses), Test Group C (4min PBM therapy + DIMS lenses), and Control Group D (DIMS lenses alone)] to see if the combined therapy has similar or better myopia control effects and comparable safety, and to identify the optimal intervention duration.

Participants will:

Complete screening examinations (axial length, refractive error, visual acuity, IOP, fundus photography, OCT, etc.) and sign the informed consent form.

Be randomly assigned to one of the four groups and receive the corresponding intervention (use the Yingtong Vision Rehabilitation Instrument as per group-specific duration twice a day, with ≥4-hour interval, plus DIMS lenses; or only DIMS lenses).

Attend regular follow-up visits at 30 days, 3 months, 6 months, 9 months, and 12 months for efficacy and safety assessments (including repeated ocular examinations and adverse event reporting).

Cooperate with the entire 12-month trial process and comply with the device usage specifications and follow-up requirements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 14 years old, regardless of gender;
* After cycloplegic autorefraction, monocular or binocular spherical equivalent refraction (SER) meets: -6.00D ≤ SER ≤ -1.00D, and binocular best-corrected visual acuity (BCVA) ≥ 0.8 (logMAR 0.1; Snellen 20/25);
* Binocular anisometropia ≤ 1.50D; astigmatism ≤ 2.50D;
* Able to understand the purpose of the study, willing to participate in this clinical verification, sign the informed consent form personally or through their legal guardian, and cooperate with the entire trial process (12 months).

Exclusion Criteria:

* Photophobia or allergy to cycloplegic agents (e.g., tropicamide or cyclopentolate);
* Received any of the following myopia control measures within one month (including but not limited to): low-concentration atropine eye drops, orthokeratology lenses, myopia control-related frame glasses, low-level red light therapy, defocus soft contact lenses, or defocus RGP lenses;
* Subjects with ocular diseases that may affect visual acuity or refractive error (e.g., lens disorders such as cataracts, glaucoma, macular degeneration, corneal diseases, uveitis, retinal detachment, severe vitreous opacity, etc.);
* Neurological diseases (previous convulsion history, epilepsy, tic disorders, central nervous system developmental abnormalities) or mental and psychological diseases;
* Systemic diseases: immune system diseases, central nervous system diseases, Down syndrome, asthma, severe cardiopulmonary function impairment, severe liver and kidney dysfunction, acute or chronic sinusitis, or diabetes mellitus;
* Binocular manifest strabismus or any other pathological changes of the eyeball or acute inflammatory ocular diseases;
* Subjects deemed inappropriate by the investigator.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 364 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
6-month axial length change | 6-month
  The difference in axial length at 6 months after trial initiation compared with the baseline axial length

SECONDARY OUTCOMES:
1-, 3-, 9- and 12-month axial length changes | 1-, 3-, 9- and 12-month
  The difference in axial length at 1-, 3-, 9- and 12-month after trial initiation compared with the baseline axial length
12-month spherical equivalent refraction (SER) change | 12-month
  The difference in spherical equivalent refraction at 12-month after trial initiation compared with the baseline spherical equivalent refraction

OTHER OUTCOMES:
Adverse event rate and serious adverse event rate | 1-, 3-, 6-, 9- and 12-month
  Adverse event rate and serious adverse event rate
12-month visual adverse event rate | 12-month
  BVCA decrease ≥0.2 logMAR

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second People's Hospital of Foshan City, Foshan, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Fourth People's Hospital of Shenyang City, Shenyang, Liaoning
  - The First Affiliated Hospital of Guangxi Medical University, Guilin, Nanning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Result] Zhao J, Pan X, Sui R, Munoz SR, Sperduto RD, Ellwein LB. Refractive Error Study in Children: results from Shunyi District, China. Am J Ophthalmol. 2000 Apr;129(4):427-35. doi: 10.1016/s0002-9394(99)00452-3. PMID 10764849
- [Result] Maul E, Barroso S, Munoz SR, Sperduto RD, Ellwein LB. Refractive Error Study in Children: results from La Florida, Chile. Am J Ophthalmol. 2000 Apr;129(4):445-54. doi: 10.1016/s0002-9394(99)00454-7. PMID 10764851
- [Result] Pokharel GP, Negrel AD, Munoz SR, Ellwein LB. Refractive Error Study in Children: results from Mechi Zone, Nepal. Am J Ophthalmol. 2000 Apr;129(4):436-44. doi: 10.1016/s0002-9394(99)00453-5. PMID 10764850
- [Result] Mutti DO, Hayes JR, Mitchell GL, Jones LA, Moeschberger ML, Cotter SA, Kleinstein RN, Manny RE, Twelker JD, Zadnik K; CLEERE Study Group. Refractive error, axial length, and relative peripheral refractive error before and after the onset of myopia. Invest Ophthalmol Vis Sci. 2007 Jun;48(6):2510-9. doi: 10.1167/iovs.06-0562. PMID 17525178
- [Result] Zadnik K, Sinnott LT, Cotter SA, Jones-Jordan LA, Kleinstein RN, Manny RE, Twelker JD, Mutti DO; Collaborative Longitudinal Evaluation of Ethnicity and Refractive Error (CLEERE) Study Group. Prediction of Juvenile-Onset Myopia. JAMA Ophthalmol. 2015 Jun;133(6):683-9. doi: 10.1001/jamaophthalmol.2015.0471. PMID 25837970
- [Result] Zhang M, Gazzard G, Fu Z, Li L, Chen B, Saw SM, Congdon N. Validating the accuracy of a model to predict the onset of myopia in children. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5836-41. doi: 10.1167/iovs.10-5592. PMID 21330664
- [Result] Jones-Jordan LA, Sinnott LT, Manny RE, Cotter SA, Kleinstein RN, Mutti DO, Twelker JD, Zadnik K; Collaborative Longitudinal Evaluation of Ethnicity and Refractive Error (CLEERE) Study Group. Early childhood refractive error and parental history of myopia as predictors of myopia. Invest Ophthalmol Vis Sci. 2010 Jan;51(1):115-21. doi: 10.1167/iovs.08-3210. Epub 2009 Sep 8. PMID 19737876
- [Result] Tedja MS, Wojciechowski R, Hysi PG, Eriksson N, Furlotte NA, Verhoeven VJM, Iglesias AI, Meester-Smoor MA, Tompson SW, Fan Q, Khawaja AP, Cheng CY, Hohn R, Yamashiro K, Wenocur A, Grazal C, Haller T, Metspalu A, Wedenoja J, Jonas JB, Wang YX, Xie J, Mitchell P, Foster PJ, Klein BEK, Klein R, Paterson AD, Hosseini SM, Shah RL, Williams C, Teo YY, Tham YC, Gupta P, Zhao W, Shi Y, Saw WY, Tai ES, Sim XL, Huffman JE, Polasek O, Hayward C, Bencic G, Rudan I, Wilson JF; CREAM Consortium; 23andMe Research Team; UK Biobank Eye and Vision Consortium; Joshi PK, Tsujikawa A, Matsuda F, Whisenhunt KN, Zeller T, van der Spek PJ, Haak R, Meijers-Heijboer H, van Leeuwen EM, Iyengar SK, Lass JH, Hofman A, Rivadeneira F, Uitterlinden AG, Vingerling JR, Lehtimaki T, Raitakari OT, Biino G, Concas MP, Schwantes-An TH, Igo RP Jr, Cuellar-Partida G, Martin NG, Craig JE, Gharahkhani P, Williams KM, Nag A, Rahi JS, Cumberland PM, Delcourt C, Bellenguez C, Ried JS, Bergen AA, Meitinger T, Gieger C, Wong TY, Hewitt AW, Mackey DA, Simpson CL, Pfeiffer N, Parssinen O, Baird PN, Vitart V, Amin N, van Duijn CM, Bailey-Wilson JE, Young TL, Saw SM, Stambolian D, MacGregor S, Guggenheim JA, Tung JY, Hammond CJ, Klaver CCW. Genome-wide association meta-analysis highlights light-induced signaling as a driver for refractive error. Nat Genet. 2018 Jun;50(6):834-848. doi: 10.1038/s41588-018-0127-7. Epub 2018 May 28. PMID 29808027
- [Result] Wang W, Jiang Y, Zhu Z, Zhang S, Xuan M, Chen Y, Xiong R, Bulloch G, Zeng J, Morgan IG, He M. Clinically Significant Axial Shortening in Myopic Children After Repeated Low-Level Red Light Therapy: A Retrospective Multicenter Analysis. Ophthalmol Ther. 2023 Apr;12(2):999-1011. doi: 10.1007/s40123-022-00644-2. Epub 2023 Jan 7. PMID 36609829
- [Result] Boyer D, Hu A, Warrow D, Xavier S, Gonzalez V, Lad E, Rosen RB, Do D, Schneiderman T, Ho A, Munk MR, Jaffe G, Tedford SE, Croissant CL, Walker M, Ruckert R, Tedford CE. LIGHTSITE III: 13-Month Efficacy and Safety Evaluation of Multiwavelength Photobiomodulation in Nonexudative (Dry) Age-Related Macular Degeneration Using the Lumithera Valeda Light Delivery System. Retina. 2024 Mar 1;44(3):487-497. doi: 10.1097/IAE.0000000000003980. PMID 37972955
- [Result] Ivandic BT, Ivandic T. Low-level laser therapy improves visual acuity in adolescent and adult patients with amblyopia. Photomed Laser Surg. 2012 Mar;30(3):167-71. doi: 10.1089/pho.2011.3089. Epub 2012 Jan 11. PMID 22235969
- [Result] Kaymak H, Munk MR, Tedford SE, Croissant CL, Tedford CE, Ruckert R, Schwahn H. Non-Invasive Treatment of Early Diabetic Macular Edema by Multiwavelength Photobiomodulation with the Valeda Light Delivery System. Clin Ophthalmol. 2023 Nov 22;17:3549-3559. doi: 10.2147/OPTH.S415883. eCollection 2023. PMID 38026594
- [Result] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681
- [Result] Linnik LA, Usov NI, Chechin PP, Pelepchuk OS. [Prospects for using stimulating laser therapy in ophthalmology]. Oftalmol Zh. 1982;37(4):193-7. No abstract available. Russian. PMID 7145299
- [Result] Posten W, Wrone DA, Dover JS, Arndt KA, Silapunt S, Alam M. Low-level laser therapy for wound healing: mechanism and efficacy. Dermatol Surg. 2005 Mar;31(3):334-40. doi: 10.1111/j.1524-4725.2005.31086. PMID 15841638
- [Result] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT07330180/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT07330180/ICF_001.pdf